CLINICAL TRIAL: NCT02811588
Title: Registry of Stable Hypercapnic Chronic Obstructive Pulmonary Disease Treated With Non-Invasive Ventilation Amendment: Home Tele-Monitoring of Non-Invasive Ventilation in Chronic Obstructive Pulmonary Disease
Brief Title: HomeVent ( Connect) Registry: EU COPD Home NIV Registry
Acronym: HOmeVent
Status: Active, not recruiting | Type: Observational
Sponsor: ResMed (Industry)
Collaborators: CRI-The Clinical Research Institute GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: CA5 - NIV COPD Registry EU
Record Dates: First submitted 2016-06-09; First posted 2016-06-23 (Estimated); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Noninvasive Ventilation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Phase1:Screening phase: normocapnic group: Normocapnic COPD patients
- Phase1;Screening phase: hypercapnic group: Hypercapnic COPD patients
- Phase1:Treatment phase: control group: Hypercapnic COPD patients in whom NIV is not indicated or who have contraindication(s) for, or refuse, NIV treatment.
- Phase1:Treatment phase: non-invasive ventilation group: Hypercapnic COPD patients in whom NIV is indicated and who accept NIV treatment.
  Interventions: Device: Non-invasive ventilation

INTERVENTIONS:
Device: Non-invasive ventilation
  Groups: Phase1:Treatment phase: non-invasive ventilation group

SUMMARY:
The prevalence of chronic respiratory disease, including chronic obstructive pulmonary disease (COPD), is increasing in industrialized countries. Over the next decade deaths from COPD are projected to increase by more than 30% and COPD will become the third leading cause of death worldwide by 2030. There is robust scientific evidence that non-invasive ventilation (NIV) therapy is an effective option for most COPD patients hospitalized with acute hypercapnic respiratory failure secondary to an acute disease exacerbation. More recently, NIV has been shown to significantly improve survival and quality of life in COPD patients with chronic stable hypercapnic disease. These data represent an important advance in the field, and indicate that usage of NIV in patients with chronic stable hypercapnic COPD should increase. Such an increase would be expected to improve patient outcomes and have a beneficial impact on the significant healthcare burden incurred by these patients. However, the proportion of stable COPD patients with chronic hypercapnia is unknown. In addition, using NIV at home to treat COPD patients with hypercapnic (type 2) respiratory failure has not often been considered previously and there is a paucity of data regarding NIV usage patterns over time in this setting.

Phase2:

There is robust scientific evidence that non-invasive ventilation (NIV) therapy is an effective option for most COPD patients hospitalised with acute hypercapnic respiratory failure secondary to an acute disease exacerbation [3]. More recently, NIV has been shown to significantly improve survival and quality of life in COPD patients with chronic stable hypercapnic disease [4] and in patients with persistent hypercapnia after an acute chronic respiratory failure [11]. Over the past two decades, the utilisation of NIV has become one of the most important developments in the field of mechanical ventilation. However, unsuccessful NIV was found to be independently associated with death [5] and poor NIV compliance was associated with higher risk of repeat acute NIV use [6]. There is a paucity of useful predictors of poor patient compliance and the performance of conventional algorithms for detecting COPD exacerbations is still weak. Detection of NIV failure is crucial in patient management in view of its negative effect on quality of life and prognosis and the fact that it often leads to hospitalisation. In addition, 70% of COPD-related healthcare costs are consequences of emergency and hospital stays for the treatment of exacerbations [7].

Recently, tele-monitoring emerged and unfolded differently among various healthcare organisations and countries. Evidence regarding its impact on the management of COPD patients is still insufficient to draw firm conclusions. Assumption has been made that remote monitoring of home NIV treatment could help to identify novel predictors of the early detection of NIV failure and deteriorations in patients with COPD. The incidence in routine clinical care of unplanned all-cause and COPD-caused hospitalisations in patients treated with NIV therapy who are continuously monitored by telemetric data in several European countries needs evaluation. In addition, predictors of unplanned all-cause and COPD-caused hospitalisations as well as of compliance and persistence to NIV therapy should be assessed in this patient population with special respect to continuous tele-monitoring

DETAILED DESCRIPTION:
Pre-Screening and check of eligibility Routine clinical care patients are diagnosed and checked for potential eligibility of study participation based on existing data generated in routine clinical care which is not part of this observational study Prescription of treatment The decision of prescription of NIV therapy to the individual patient lies with the treating physician during the course of routine clinical care and is not part of this observational study. Diagnosis of COPD and indication of NIV therapy as well as initiation of treatment should follow applicable medical guidelines and local clinical care policy. Prescription and use of adequate ResMed NIV devices with tele-monitoring option according to Annex 1, 3. have to follow the current instructions for use (IFU) of each device.

Screening and enrolment visit Patients will be screened and enrolled by contracted study sites only, i.e. NIV expert centres.

Screening of potentially eligible patients will be performed within routine clinical care using data created within routine clinical care. Adequate staff members of the study site will inform potentially eligible patients about the potential use of their medical and telemetric data within this observational study by information documents which have been approved by the responsible Ethics Committee. Within this study medical care of the patient is not in any way touched by protocol definitions but an individual decision by the treating physician in routine clinical care. Only use and handling of medical and telemetric data for scientific purposes defined in this protocol are elements of informed consent. The patient will be given sufficient time to consider informed consent to data handling and to get answers to his questions. If the patient agrees, the informed consent form for data use will be provided for signature.

After patients' signing, patients are screened and checked for eligibility according to in- and exclusion criteria by the participating sites, either on every day consecutively or at pre-defined schedules (e.g. on defined days of the week, only) to minimise selection bias. Medical screening includes check of COPD according to medical guidelines.

Study relevant data will be reported in the e-CRF. The system will automatically display the patient ID as consecutive number across all participating study sites, i.e. without reference to the recruiting site.

The following data items will be documented of each participating patient:

Demographic data Patient's physical status Patient's social status Medical history Concomitant medication and diseases Data regarding COPD diagnosis Spirometry results (no older than 1 month) Blood gas analyses (carbon dioxide and bicarbonate concentration) during spontaneous breathing (pH>7.35) at date of decision making on initiation of NIV therapy Date of NIV therapy prescription Telemetric data of NIV device settings will be recorded as soon as the device has been delivered to the patient and was used for the first time Amount of supplemental oxygen during NIV (if needed) The patients will further be asked to answer the SRI questionnaire (refer to Annex 2), and the CAT questionnaire Initiation of treatment Initiation of NIV therapy (the device has been delivered to the patient and was used for the first time) after prescription should start according to local routine clinical care before or as soon as possible after enrolment into the study (with a maximum of 7 days before enrolment). Current medical guidelines and recommendations apply, however, they might differ in participating countries, and thus, prescription and initiation of NIV therapy is the decision of the treating physician and will follow local policies. Data on initiation of NIV therapy will be recorded by telemetric data as soon as the device has been delivered to the patient and was used for the first time.

Follow-up visits In routine clinical care, a first control visit of the patient at the site after NIV therapy initiation should take place within the first 6 months together with nocturnal assessment of ventilator therapy [12]. It is recommended that subsequent control visits at the site should be performed at least 1-2 times a year [12]. To ensure comparability of FU data, at least one follow-up visit at the site within 12 months of follow-up should be performed (if in line with routine clinical care).

At the FU visit at the site the following data from routine clinical care data should be documented in the e-CRF:

Patient status Concomitant medication and diseases Spirometry results (no older than 3 months) Body plethysmography (if available) Blood gas analyses (carbon dioxide, pH and bicarbonate concentration) during spontaneous breathing Serious adverse events since last site visit. History of exacerbations not leading to a hospitalisation The patient will again be asked to answer to the SRI and CAT questionnaires. NIV device settings and other device data will continuously be transferred in FU as tele-monitoring data.

Follow-up questionnaires Every six months of follow-up short questionnaires asking for hospitalisations and other potential SAEs since last contact will be sent by mail to all patients. Closed envelopes with PID outside including the questionnaire and a free return envelope will be prepared and sent to site by the CRO. Site staff will forward the envelope to the corresponding patient who is asked to return the completed questionnaire (which contains pseudonymous data only) directly to CRI using the free reply envelope. In case of missing answer after one written reminder the study site should contact the patient by phone in order to obtain the required information.

Data regarding hospitalisations or SAEs reported by the patient will be documented in the e-CRF primarily by the CRO on the basis of available medical data. In case a patient reports a hospitalisation or other SAE, the responsible study site will be informed by the CRO and will subsequently contact the patient's family doctor respectively the hospital where the patient was treated and ask for supportive documents (i.e. hospital discharge letter, diagnostic reports) as applicable. The study site is subsequently responsible for completion of event data.

These procedures will not be performed in study patients enrolled in the ANTADIR registry in France and used for joined analysis in this study. Thus, analysis of hospitalisations will therefore be performed for patients enroled in Germany, Spain, UK and other potentially participating countries but not for patients

ELIGIBILITY:
Phase1:Inclusion Criteria:

* Age ≥18 years
* GOLD stage 3 or 4 COPD
* pCO2 value available not older than one month
* Ability to fully understand the study information and willing to give informed consent

Phase2:

Age ≥18 years COPD eligible for NIV treatment (according to applicable medical guidelines and local policy in routine clinical care) Prescription of an adequate ResMed NIV device with tele-monitoring option (according to Annex 1, 3.) as part of routine clinical care Acceptance of tele-monitoring and corresponding data handling Naive to long-term NIV treatment with initiation of NIV either ≤7 days before or after enrolment into study Able to fully understand information on data protection and provide written informed consent for use of corresponding medical and telemetric data.

Phase1:Exclusion Criteria:Existing treatment with NIV Phase2:Exclusion Criteria Invasive ventilation therapy Another life-threatening disease with estimated survival < 12 months (other than COPD, e.g. cancer) Further exclusion criteria according to IFU of the device intended and prescribed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately 550 adult female and male patients with COPD eligible for NIV treatment will be enrolled, out of which 231 patients have been enrolled within the phase 1 of the study. If a patient is enrolled into the study but is never using the prescribed device (i.e. refusal of prescribed therapy) he/she will be replaced.
  If a patient, who has already started NIV therapy, is enrolled, the start of therapy must not be longer than 7 days before enrolment.
  Within this study population, data of a maximum of about 100 patients will be added by the French ANTADIR registry in line with in- and exclusion criteria of this observational study.
Sampling Method: Non-Probability Sample
Enrollment: 169 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Phase 1: Prevalence of hypercapnia in patients with GOLD stage 3 and 4 COPD. | Phase1:July 2017
Phase2:Incidence of unplanned all-cause hospitalisations in routine clinical care in patients treated with NIV therapy who are continuously monitored by telemetric data | Dec20-Dec22
  Unplanned hospitalisation is within this protocol defined as ill-defined hospital admissions in acute inpatient medical settings for any cause for more than one calendar day (overnight stay) where managing demand for unplanned admissions is a priority [13].

SECONDARY OUTCOMES:
Patterns of NIV use | July 2017
  Device reported NIV usage
Phase2:Incidence of unplanned COPD-caused hospitalisations | Dec20-Dec22
  COPD-caused hospitalisation is within this protocol defined as COPD exacerbation leading to hospitalisation as defined above.
Phase2:Predictors of unplanned all-cause hospitalisations | Dec20-Dec22
  Hospitalisation is within this protocol defined as inpatient care of more than one calendar day (overnight stay) for any cause. Overnight survey visits (e.g. sleep lab) are not considered "hospitalisation".
Phase2:Predictors of unplanned COPD-caused hospitalisations | Dec20-Dec22
  COPD-caused hospitalisation is within this protocol defined as COPD exacerbation leading to hospitalisation as defined above.
Phase2:Predictors of compliance and persistence to NIV therapy | Dec20-Dec22

CONTACTS AND LOCATIONS:
Overall Officials: Michael Dreher, Prof, Principal Investigator — University Hospital, Aachen; Nicholas Hart, Prof, Study Chair — NHS Foundation; Claudio Rabec, Prof, Study Chair — Centre Hospitalier et Universitaire Dijon
Locations (4):
- Germany (4):
  - Universitätsklinikum Aachen, Aachen, North Rhine-Westphalia
  - Clemenshospital, Münster, Westfalen Lippe
  - Marienkrankenhaus gGmbH, Soest, Westfalen Lippe
  - Kliniken der Stadt Köln, Cologne

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mannino DM, Buist AS. Global burden of COPD: risk factors, prevalence, and future trends. Lancet. 2007 Sep 1;370(9589):765-73. doi: 10.1016/S0140-6736(07)61380-4. PMID 17765526
- [Background] Brochard L, Mancebo J, Wysocki M, Lofaso F, Conti G, Rauss A, Simonneau G, Benito S, Gasparetto A, Lemaire F, et al. Noninvasive ventilation for acute exacerbations of chronic obstructive pulmonary disease. N Engl J Med. 1995 Sep 28;333(13):817-22. doi: 10.1056/NEJM199509283331301. PMID 7651472
- [Result] Dreher M, Neuzeret PC, Windisch W, Martens D, Hoheisel G, Groschel A, Woehrle H, Fetsch T, Graml A, Kohnlein T. Prevalence Of Chronic Hypercapnia In Severe Chronic Obstructive Pulmonary Disease: Data From The HOmeVent Registry. Int J Chron Obstruct Pulmon Dis. 2019 Oct 18;14:2377-2384. doi: 10.2147/COPD.S222803. eCollection 2019. PMID 31695357
- See also: Global Initiative for Chronic Obstructive Lung Disease webpage — https://goldcopd.org/gold-reports/

DOCUMENTS (1):
  • Study Protocol (2020-10-01): https://cdn.clinicaltrials.gov/large-docs/88/NCT02811588/Prot_000.pdf